CLINICAL TRIAL: NCT00234078
Title: Dose-response Study of OPC-12759 Ophthalmic Suspension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 037E-04-002; JapicCTI-050040
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-01

CONDITIONS: Dry Eye Syndromes
Keywords: OPC-12759; Dry eye syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — rebamipide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.5% OPC-12759 (Experimental): 0.5% OPC-12759 (rebamipide) ophthalmic suspension
  Interventions: Drug: 0.5% OPC-12759
- 1% OPC-12759 (Experimental): 1% OPC-12759 (rebamipide) ophthalmic suspension
  Interventions: Drug: 1% OPC-12759
- 2% OPC-12759 (Experimental): 2% OPC-12759 (rebamipide) ophthalmic suspension
  Interventions: Drug: 2% OPC-12759
- placebo (Placebo Comparator): placebo of OPC-12759 (rebamipide) ophthalmic suspension
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 0.5% OPC-12759
  Arms: 0.5% OPC-12759
Drug: 1% OPC-12759
  Arms: 1% OPC-12759
Drug: 2% OPC-12759
  Arms: 2% OPC-12759
Drug: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the dose-response of OPC-12759 ophthalmic suspension in dry eye patients.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient.
2. Subjective complaint of dry eye that has been present for minimum 20 months.
3. Primary ocular discomfort severity is moderate to severe.
4. Corneal - conjunctival damage is moderate to severe.
5. Unanesthetized Schirmer's test score of 7mm/5minutes or less.
6. Best corrected visual acuity of 0.2 or better in both eyes.

Exclusion Criteria:

1. Presence of anterior segment disease or disorder other than that associated with keratoconjunctivitis sicca.
2. Anticipated use of any topically-instilled ocular medications or patients with cannot discontinue the use during the study.
3. Anticipated use of contact lens during the study.
4. Any history of ocular surgery within 12 months.
5. Female patients who are pregnant, possibly pregnant or breast feeding;
6. Known hypersensitivity to any component of the study drug or procedural medications.
7. Receipt of any investigational product within 4 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2005-01; Primary Completion 2006-04 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Satoshi Oshima, Study Director — Dermatologicals & Ophthalmologicals Division
Locations (1):
- Otsuka Pharmaceutical Co., Ltd., Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.5% OPC-12759: 0.5% rebamipide ophthalmic suspension received one drop of to both eyes four times a day for 12 weeks
- 1% OPC-12759: 1% rebamipide ophthalmic suspension received one drop of to both eyes four times a day for 12 weeks
- 2% OPC-12759: 2% rebamipide ophthalmic suspension received one drop of to both eyes four times a day for 12 weeks
- Placebo: 0% rebamipide ophthalmic suspension received one drop of to both eyes four times a day for 12 weeks
Period: Overall Study
Arm/Group | 0.5% OPC-12759 | 1% OPC-12759 | 2% OPC-12759 | Placebo
Started | 72 | 72 | 74 | 72
Completed | 66 | 63 | 64 | 68
Not Completed | 6 | 9 | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5% OPC-12759 | 1% OPC-12759 | 2% OPC-12759 | Placebo | Total
Number analyzed (Participants) | 72 | 72 | 74 | 72 | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (13.6) | 62.5 (13.5) | 60.3 (11.5) | 56.0 (16.2) | 59.8 (13.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 38 | 47 | 45 | 169
  >=65 years | 33 | 34 | 27 | 27 | 121
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 65 | 70 | 65 | 266
  Male | 6 | 7 | 4 | 7 | 24
Region of Enrollment [Number; unit: participants]
  Japan | 72 | 72 | 74 | 72 | 290

OUTCOME MEASURES:

1. Primary Outcome: Change in Fluorescein Corneal Staining (FCS) Score From Baseline to Last Observation Carried Forward (LOCF)
Description: FCS indicates the damage to the corneal epithelium. Per the National Eye Institute/Industry Workshop report, the cornea was divided into 5 fractions, each of which was given a staining score from 0 to 3, and the total score was calculated (0-15). 0 is better. The change from baseline (CFB) to LOCF at the end of instillation (LOCF endpoint) was used to analyze dose-response. A general linear model was used to examine if slope parameters were not equal to zero.
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 0.5% OPC-12759 | 1% OPC-12759 | 2% OPC-12759 | Placebo
Number analyzed (Participants) | 72 | 72 | 74 | 72
scores on a scale | -2.8 (2.3) | -3.1 (2.6) | -2.1 (2.8) | -2.6 (2.7)
Statistical Analysis 1: Comparison: 0.5% OPC-12759 vs 1% OPC-12759 vs 2% OPC-12759 vs Placebo; Test type: Superiority or Other; p = 0.385, t-test, 2 sided — versus placebo; a general linear model

2. Primary Outcome: Change in Primary Ocular Discomfort (POD) Score From Baseline to Last Observation Carried Forward (LOCF)
Description: POD indicates the ocular symptom most bothersome to the patient. POD selected by each patient from among the following ocular symptoms; Foreign body sensation, Dryness, Photophobia, Eye pain and Blurred vision. POD was scored from 0 through 4; a score of 0 indicated no symptoms and a score of 4 indicated very severe symptoms. 0 is better. The change from baseline (CFB) to LOCF at the end of instillation (LOCF endpoint) was used to analyze dose-response. A general linear model was used to examine if slope parameters were not equal to zero.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 0.5% OPC-12759 | 1% OPC-12759 | 2% OPC-12759 | Placebo
Number analyzed (Participants) | 72 | 72 | 74 | 74
scores on a scale | -1.2 (1.1) | -1.4 (1.0) | -1.3 (1.1) | -1.3 (0.9)
Statistical Analysis 1: Comparison: 0.5% OPC-12759 vs 1% OPC-12759 vs 2% OPC-12759 vs Placebo; Test type: Superiority or Other; p = 0.601, t-test, 2 sided — versus placebo; a general linear model

3. Post Hoc Outcome: Change in Fluorescein Corneal Staining (FCS) Score From Baseline to Week 12
Description: FCS indicates the damage to the corneal epithelium. Per the National Eye Institute/Industry Workshop report, the cornea was divided into 5 fractions, each of which was given a staining score from 0 to 3, and the total score was calculated (0-15). 0 is better. The CFB in the FCS scores were compared between the 0.5, 1 and 2% rebamipide group and the placebo group using a Dunnett's t-test
Time Frame: Baseline, 12week
Population: From the FAS of 290 patients, 218 patients who had no punctal plug insertion or punctal occlusion and who had a baseline schirmer test value of equal to or less than 5 mm for the eye evaluated for efficacy were selected and subjected to exploratory data analysis
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 0.5% OPC-12759 | 1% OPC-12759 | 2% OPC-12759 | Placebo
Number analyzed (Participants) | 56 | 50 | 46 | 51
scores on a scale | -3.2 (2.1) | -3.5 (2.4) | -2.9 (2.5) | -2.2 (2.6)
Statistical Analysis 1: Comparison: 0.5% OPC-12759 vs Placebo; Test type: Superiority or Other; p = 0.084, t-test, 2 sided — p-value is adjusted for multiple comparisons
Statistical Analysis 2: Comparison: 1% OPC-12759 vs Placebo; Test type: Superiority or Other; p = 0.020, t-test, 2 sided — p-value is adjusted for multiple comparisons
Statistical Analysis 3: Comparison: 2% OPC-12759 vs Placebo; Test type: Superiority or Other; p = 0.421, t-test, 2 sided — p-value is adjusted for multiple comparisons

4. Post Hoc Outcome: Change in Lissamine Green Conjunctival Staining (LGCS) Score From Baseline to Week 12
Description: LGCS indicates the damage to the conjunctival epithelium. Per the National Eye Institute/Industry Workshop report, the conjunctiva was divided into 6 fractions, each of which was given a staining score from 0 to 3, and the total score was calculated (0-18). 0 is better. The CFB in the LGCS scores were compared between the 0.5, 1 and 2% rebamipide group and the placebo group using a Dunnett's t-test.
Time Frame: Baseline, 12weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 0.5% OPC-12759 | 1% OPC-12759 | 2% OPC-12759 | Placebo
Number analyzed (Participants) | 56 | 50 | 46 | 51
scores on a scale | -3.8 (3.1) | -4.5 (3.3) | -4.2 (3.2) | -2.5 (3.2)
Statistical Analysis 1: Comparison: 0.5% OPC-12759 vs Placebo; Test type: Superiority or Other; p = 0.087, t-test, 2 sided — p-value is adjusted for multiple comparisons
Statistical Analysis 2: Comparison: 1% OPC-12759 vs Placebo; Test type: Superiority or Other; p = 0.004, t-test, 2 sided — p-value is adjusted for multiple comparisons
Statistical Analysis 3: Comparison: 2% OPC-12759 vs Placebo; Test type: Superiority or Other; p = 0.029, t-test, 2 sided — p-value is adjusted for multiple comparisons

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | 0.5% OPC-12759 | 1% OPC-12759 | 2% OPC-12759 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/72 | 0/72 | 2/74 | 2/72
Other Adverse Events (participants affected / at risk) | 32/72 | 29/72 | 43/74 | 23/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5% OPC-12759 (N=72) | 1% OPC-12759 (N=72) | 2% OPC-12759 (N=74) | Placebo (N=72)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5% OPC-12759 (N=72) | 1% OPC-12759 (N=72) | 2% OPC-12759 (N=74) | Placebo (N=72)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Eye discharge (Eye disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
Eye irritation (Eye disorders) | 4 (4) | 2 (2) | 3 (3) | 3 (3)
Eye pain (Eye disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2)
Eye pruritus (Eye disorders) | 6 (6) | 4 (4) | 4 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 15 (15) | 14 (14) | 13 (13) | 17 (17)
Blood cholesterol increased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Dysgeusia (bitter taste) (Nervous system disorders) | 11 (11) | 15 (15) | 19 (19) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No